CLINICAL TRIAL: NCT00695136
Title: An Investigation of the Relationship Between Donepezil Enhanced REM Sleep, Sleep Architecture and Behavior in the Prepubertal Child With Autism
Brief Title: The Effect of Donepezil (Aricept(Registered Trademark)) on REM Sleep in Children With Autism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Swedo, M.D., Chief, Pediatrics & Developmental Neuroscience Branch, NIMH, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 080154; 08-M-0154 (Other: NIH Protocol Number)
Record Dates: First submitted 2008-06-10; First posted 2008-06-11 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Autism; Cognition Disorder
Keywords: Autism; Cognitive Disorder; Sleep; Autism Spectrum Disorder; ASD
MeSH Terms: conditions — Autistic Disorder; Cognition Disorders; Cognitive Dysfunction; Autism Spectrum Disorder | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label single arm (Experimental): Single group study of Donepezil
  Interventions: Drug: Donepezil hydrochloride; Behavioral: Increase REM sleep percentage

INTERVENTIONS:
Drug: Donepezil hydrochloride
Behavioral: Increase REM sleep percentage

SUMMARY:
This study will test whether donepezil (Aricept(Registered Trademark)), a drug that is approved by the Food and Drug Administration to treat Alzheimer's disease, can increase rapid eye movement (REM) sleep in children with autism and autism spectrum disorder (ASD). Some children with autism and ASD spend very little time in REM sleep. In some studies, decreased REM sleep has been associated with learning and behavior problems. Donepezil can increase REM sleep in some adults with different disorders. If it can increase REM sleep in children in this study, it might be able to be used in future studies to see if it can help learning and behavior problems in children with autism and ASD.

Children between 2 and 10 years of age with autism or an ASD whose percentage of REM sleep time is well below the average for children of the same age may be eligible for this study. Candidates are screened with a medical history, physical and neurological examinations, blood tests, electroencephalogram (EEG) and a sleep study. The sleep study requires an overnight stay at the NIH Clinical Center in which the child is monitored with electrodes for EEG and heartbeat recording, a tube taped below the nose to measure airflow, a probe on a finger to record oxygen levels and a small watch-like machine on the wrist to record movements.

Participating children may be required to have up to six overnight stays for sleep studies at the Clinical Center. The children start by taking 1.25 mg of donepezil for 2 to 4 weeks. Then they are admitted to the NIH Clinical Center for a sleep study, blood tests and EKG. Those whose REM sleep increases to normal levels stay on 1.25 mg of donepezil for 8 more weeks, after which they are admitted to the Clinical Center for a final physical examination, blood draw and sleep study. That ends their participation in the study.

Children whose REM sleep does not increase to normal on 1.25 mg of donepezil are given a higher dose (2.5 mg) for 2 to 4 weeks, and the above procedure is repeated. Those whose REM sleep does not increase to normal on 2.5 mg of donepezil take 5 mg of the drug for 2 to 4 weeks, and the above procedure is repeated once more. Children whose REM sleep does not increase to normal on 5 mg of donepezil stop the medication and end their participation in the study.

At each study visit, study researchers talk to the parents and examine the children to determine if donepezil is affecting the child's behavior and if the child is hav...

DETAILED DESCRIPTION:
Autism spectrum disorders are defined by aberrant development of communication and socialization in the presence of restrictive and/or repetitive behaviors. Recent epidemiologic studies have documented an increase in the number of children identified with autism spectrum disorder over the past decade and according to some, the current numbers indicate a prevalence of 1 per 150 (CDC, MMWR 2007, Feb 9th release). Despite the pressing need to identify causal factors, etiology remains elusive. Furthermore, the heterogeneity of presentation complicates attempts to locate autism's home in the brain.

Polysomnography is a reliable non-invasive tool that can be used to study the basic pathophysiological mechanisms of autism and other developmental and neuropsychiatric disabilities. Our preliminary data in young children with autism supports a growing body of literature demonstrating that sleep architecture is abnormal in this disorder. Previous studies in children with autism have identified various abnormalities in REM sleep including the following: immature organization, decreased quantity, abnormal twitches, undifferentiated sleep and REM sleep behavior disorder characterized by the absence of the muscle atonia that is normal in REM sleep and resulting in an acting out of dreams phenomenon (Tanguay et al ,.1976, Elia et al., 2000, Diomedi et al. 1999, and Thirumalai et al., 2002).

Our cohort spent an abnormally short time in the REM sleep stage of sleep compared to total sleep time (hereafter referred to as SPT REM% for REM sleep as a percent of sleep period time), and had a prolonged latency to REM sleep. The function of REM sleep and its relationship to cognition and overall neurological health is unknown and a subject of ongoing research. We know from animal studies that REM sleep increases after intensive learning sessions. These laboratory findings formed the basis for the hypothesis that this sleep stage is important for cognitive processes and that REM sleep may be useful as an indicator of brain plasticity. Current studies continue to add support for this idea. REM sleep has most recently been implicated in the process of human memory consolidation and several studies suggest that it is crucial to normal cognitive function and in the processing of emotion in memory systems. Acetylcholine (Ach) is one of the major neurotransmitters necessary for normal sleep transitions and abnormalities in Ach have been implicated in REM deficient sleep in other populations, most notably Alzheimer's disease.

This proposal is for a 6 to 20 week, single arm, open-label study to evaluate the ability of donepezil hydrochloride to enhance REM sleep in children with autism spectrum disorder found to have a low SPT REM% (defined as below 2 standard deviations of observed normative data for age). All patients will come through the screening protocol 06-M-0065. Those who meet a research diagnosis of autism spectrum disorder and are ages 2 to 11 (through the tenth year) will be evaluated for inclusion/exclusion criteria for the study.

The primary outcome measure of this protocol is to increase the SPT REM% in children with autism such that their REM/non-REM ratios begin to approach normative values. Donepezil enhanced REM sleep has been achieved in young healthy adults, in elderly, healthy adults and in elderly, demented adults with Alzeheimer's disease. Furthermore, the studies in Alzheimer disease by Mizuno et al showed a positive correlation between improved cognition and increased SPT REM %. If REM sleep is necessary for normal cognition, and its deficiency or absence can be remedied by pharmacologic intervention, then it may follow that improvement of REM sleep correlates with improved short and long term cognition in children with autism. Donepezil enhanced REM sleep has not been documented in children. Polysomnography provides a non-invasive tool to assess the effects of enhancing cholinergic tone on the abnormal sleep architecture we have documented in our pediatric, autistic population.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of autism spectrum disorder
* Male or female subjects, ages 2 through 10 years.
* Each legal guardian must have a level of understanding sufficient to agree to all required tests and examinations. Each legal guardian must understand the nature of the study.
* Each subject must be stable for at least 6 weeks on any medication or therapy regimen prior to entry into study and must have no newly (within 6 weeks) recognized or intolerable adverse effects from that medicine or therapy. No subjects will be asked to discontinue any medication in order to qualify for enrollment.

EXCLUSION CRITERIA:

* Serious, unstable illnesses including, gastroenterologic, respiratory, cardiovascular endocrinologic, immunologic,or hematologic disease.
* Renal or hepatic dysfunction that would interfere with excretion or metabolism of donepezil as evidenced by increase above upper limits of normal for BUN/creatinine, or two-fold elevation of serum transaminases (ALT/SGPT, AST/SGOT) or gamma glutamate (GGT)
* Documented history of hypersensitivity or intolerance to donepezil or other piperidine derivative.
* Subjects must not be taking any medication known to affect REM sleep or that is contraindicated for co-administration with donepezil.
* Presence or history of neurological disorders, including seizure disorders.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] McGrath MJ, Cohen DB. REM sleep facilitation of adaptive waking behavior: a review of the literature. Psychol Bull. 1978 Jan;85(1):24-57. No abstract available. PMID 203966
- [Background] Mirmiran M, van den Dungen H, Uylings HB. Sleep patterns during rearing under different environmental conditions in juvenile rats. Brain Res. 1982 Feb 11;233(2):287-98. doi: 10.1016/0006-8993(82)91203-3. PMID 7059812
- [Background] Guzman-Marin R, Ying Z, Suntsova N, Methippara M, Bashir T, Szymusiak R, Gomez-Pinilla F, McGinty D. Suppression of hippocampal plasticity-related gene expression by sleep deprivation in rats. J Physiol. 2006 Sep 15;575(Pt 3):807-19. doi: 10.1113/jphysiol.2006.115287. Epub 2006 Jul 6. PMID 16825295

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Children were screened with polysomnography and 8 of 16 subjects were found to have low REM sleep% and were eligible to continue with the study. One of the 8 elected not to participate in the dose-finding drug administration.
Groups:
- Open Label Single Arm: The children start by taking 1.25 mg of donepezil for 2 to 4 weeks. Those whose REM sleep increases to normal levels stay on 1.25 mg of donepezil for 8 more weeks. That ends their participation in the study.
  Children whose REM sleep does not increase to normal on 1.25 mg of donepezil are given a higher dose (2.5 mg) for 2 to 4 weeks. Those whose REM sleep does not increase to normal on 2.5 mg of donepezil take 5 mg of the drug for 2 to 4 weeks. Children whose REM sleep does not increase to normal on 5 mg of donepezil stop the medication and end their participation in the study.
Period: Overall Study
Arm/Group | Open Label Single Arm
Started | 7 (7)
Completed | 5
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — unrelated adverse event | 1

BASELINE CHARACTERISTICS:
Population: 16 subjects completed screening and had baseline data. However, only 8 of them were eligible for further study participation and only 5 completed the drug and provided data for analysis.
Groups:
- Open Label Single Arm: Single group study of Donepezil
  Increase REM sleep percentage :
  Donepezil hydrochloride :
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 5.08 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Time That Subjects With Autism Spend in REM Sleep.
Time Frame: 1 month (from baseline to 1.25 mg dose)
Measure: Mean (Standard Error); unit: percentage of REM sleep
Arm/Group | Open Label Single Arm
Number analyzed (Participants) | 5
percentage of REM sleep | 9.2 (2.6)

ADVERSE EVENTS:
Arm/Group | Open Label Single Arm
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Single Arm (N=7)
other (Nervous system disorders) | 1 (1) — Specific event term omitted for privacy.

LIMITATIONS AND CAVEATS:
No controls and small number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes